CLINICAL TRIAL: NCT05554757
Title: In Vivo Comparative Study of Two Different Rubber Dam System in Dental Practices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Aqsa Waheed, Principal investigator, Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AQ27101996
Record Dates: First submitted 2022-07-22; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Tooth Decay
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional rubber dam system (Experimental): in the first 30 patients, the conventional rubber dam was used prior to the OptraDam For the first 30 patients, on the day of the first appointment, the stopwatch was set for recording the time taken for the application of the conventional rubber dam . Following this, the required dental treatment was carried out. Radiographs were taken as & when necessary . At the end of the appointment, the questionnaires were filled by the patient as well as the operator regarding their experience of the conventional rubber dam
  Interventions: Device: conventional rubber dam system
- OPTRADAM (Active Comparator): In second appoinment the optradam was applied. The stopwatch was set for the recording the time of application of the OptraDam. The required dental treatment was carried out. Radiographs were taken. At the end of the appointment, the questionnaires were again filled by the patient as well as the operator regarding their experience of the OptraDam.
  Interventions: Device: OPTRADAM

INTERVENTIONS:
Device: conventional rubber dam system — rubber dam is a protective sheet with a hole that a dental professional positions over a tooth during an endodontic procedureEndodontists . This allows to isolate the treatment area with a dental clamp around the tooth. The dental sheet is placed around the in the Dental Rubber Dams and then a u-shaped device is hooked around. This isolates the single tooth where dental treatment will be conducted.
  Arms: conventional rubber dam system
Device: OPTRADAM — OptraDam Plus is a three-dimensional rubber dam that is flexible and has an anatomical shape, automatically stretched in an oral direction, an automatic hold of the device in the oral cavity is ensured.
  Arms: OPTRADAM

SUMMARY:
Isolation is essential for the successful placement of esthetic restoration to avoid any contamination of cavity with saliva ,secreation,and blood dental . This study is comparison of optradam and convetional rubberdam system.The aim of this study is to investigate which rubberdam system is better accepted by patients and dentists

DETAILED DESCRIPTION:
This is in vivo comparative study of optradam and conventional rubber dam system.For this study , two simple questionnaires were prepared.

The first questionnaire consisted of 5 questions. It enquired into the personal details of the patient, which included the name, age & gender ,the patient's previous experience of rubber dam use

1. The teeth to be isolated
2. .The type of procedure being carried out
3. The patient's comfort regarding the conventional rubber dam & the OptraDam
4. .The patient's protection regarding the conventional rubber dam & the OptraDam.
5. The patient's preference regarding the conventional rubber dam & the OptraDam The second questionnaire consisted of 7 questions. This was to be filled by the dentist operating on the respective patient. This questionnaire enquired into

1 The time taken to apply the conventional rubber dam & the OptraDam. 2 The ease with which rubber dam could be applied.The amount of retraction & access achieved during the use of each rubber dam. 3 The amount of moisture control achieved during the use of each rubber dam. 4 he ease with which radiograph could be taken. 5 The dentist's preference regarding the conventional rubber dam & OptraDam. In the first 30 patients, the conventional rubber dam was used prior to the OptraDam. In the next 30 patients, the OptraDam was used before the conventional rubber dam. This was done to prevent bias. For the first 30 patients, on the day of the first appointment, the stopwatch was set for recording the time taken for the application of the conventional rubber dam . Following this, the required dental treatment was carried out. Radiographs were taken as & when necessary . At the end of the appointment, the questionnaires were filled by the patient as well as the operator regarding their experience of the conventional rubber dam.On the next consecutive appointment, the stopwatch was set for the recording the time of application of the OptraDam. The required dental treatment was carried out. Radiographs were taken. At the end of the appointment, the questionnaires were again filled by the patient as well as the operator regarding their experience of the OptraDam. For the next set of 30 patients, the above procedure was repeated, except that, for them the OptraDam was used prior to conventional rubber dam].

DATA ANALYSIS:

All statistical analyses are performed with SPSS 13.0 . Analyses were confined to simple cross tabulations of the patients & operator . P - value was calculated using Chi-square test

& Wilcoxon test whenever required to get appropriate results

ELIGIBILITY:
Inclusion Criteria:

Patients who agree to participate in study. Patients who came for restorative and endodontic purpose . Fully erupted molars and premolars. Patient having no previous experience with rubber dam system.

Exclusion Criteria:

Grossly carious tooth with poor prognosis. Medically compromised patients. Those Patient which are uncooperative. Patients having latex allergy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-25 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Moisture control | immediately after procedure
  clinically observing tooth moisture control with optradam and coventional rubber dam system

SECONDARY OUTCOMES:
Retraction and access | immediately after procedure
  clinically observing hindrance with clasp during procedure
radiographic ease | immediately after procedure
  radiograph easily taken with rubber dam system

CONTACTS AND LOCATIONS:
Locations (1):
- Aqsa waheed, Islamabad, Islambad, Pakistan

IPD SHARING:
Plan to Share IPD: No